CLINICAL TRIAL: NCT03296137
Title: Adoptive Cell Therapy Across Cancer Diagnoses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D. Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA1720
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: immune therapy; TILs; Adoptive cell therapy
MeSH Terms: conditions — Neoplasms | interventions — Ipilimumab; Nivolumab; aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor-infiltrating Lymphocyte (TIL) Therapy with checkpoint inhibitors (Experimental)
  Interventions: Biological: Autologous tumor-infiltrating lymphocytes; Drug: Ipilimumab; Drug: Nivolumab; Drug: proleukin; Drug: Cyclophosphamide; Drug: Fludara

INTERVENTIONS:
Biological: Autologous tumor-infiltrating lymphocytes — Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion.
Drug: Ipilimumab — One treatment with ipilimumab (3 mg/kg) prior to tumor resection.
Drug: Nivolumab — 4 doses of nivolumab. Starting 2 days prior to TIL infusion and every 2 weeks hereafter.
Drug: proleukin — 2 MIE s.c. injection, after TIL infusion and continuing for 2 weeks
Drug: Cyclophosphamide — 2 doses (60 mg/kg) prior to TIL infusion
Drug: Fludara — 5 doses (25 mg/m2) prior to TIL infusion

SUMMARY:
This study will perform tumor-infiltrating lymphocyte (TIL)-based adoptive T-cell therapy in combination with checkpoint inhibition on cancer patients across all cancer diagnoses.

DETAILED DESCRIPTION:
Adoptive cell therapy (ACT) is a personalized form of immunotherapy, where lymphocytes isolated from the patient's own tumor tissue are expanded 1000-fold ex-vivo and then infused back into the patient. The lymphocytes are then able to recognize and attack remaining cancer cells. This approach has shown remarkable clinical results in several trials conducted worldwide for patients with advanced melanoma - some with durable remissions. Promising clinical results were obtained in smaller trials where patients with disparate solid tumors were treated with tumor-infiltrating lymphocytes (TILs). At Center for Cancer Immune Therapy (CCIT) at Herlev Hospital, there are currently clinical trials undergoing in ovarian and renal cancer, and internationally ACT is being tested in an increasing number of cancer diagnoses, some trials are even recruiting patients across cancer types. Studies have shown that a high intratumoral infiltration with TILs in is correlated to the general clinical outcome of the disease in virtually all solid tumors, and thus clinical trials with TIL-based ACT to different cancer diagnoses have been undertaken.

To support the TIL-mediated tumor elimination, in classical ACT protocols patients go through a highly specialized treatment regime before and after TIL infusion. This regime includes lymphodepletion with 7 days non-myeloablative chemotherapy, to provide an immunological window of opportunity for the infused TILs, and concomitant immune stimulation with interleukin-2 (IL-2). Checkpoint inhibition to support the anti-tumor activity of TILs is currently under extensive investigation in several other trials worldwide. Thus, lymphodepletion and IL-2 stimulation are well-established as supportive therapy and already an integrated part of current ACT protocols and while checkpoint inhibition is a new addition at CCIT; internationally other centers have ongoing comparable trials.

Drug-based immunotherapy in the form of checkpoint inhibitors (anti-PD-1 and anti-CTLA-4) has yielded impressive clinical results across tumor histologies. Recent results indicate that the effect of immunotherapy relies not so much on the cancer diagnoses but rather on the genomic and immunologic features of the individual patient's cancer disease. Both ACT and checkpoint inhibition work by tipping the immunological balance in favor of activation and away from suppression or avoidance by the cancer cells. Scientific evidence now show that administering anti-CTLA-4 and PD-1 could provide a benefit in the ACT setting, and several ongoing clinical trials are testing combinations of ACT and checkpoint inhibition. To synergistically maximize the immunological potential, we wish to combine ACT with an anti-CTLA-4 antibody (Ipilimumab) prior to tumor resection and an anti-PD-1 antibody (Nivolumab) in combination with TIL infusion.

Patients will be treated with one dose of Ipilimumab 14 days before undergoing surgery to harvest tumor material for TIL production. Patients is admitted on day -8 in order to undergo lymphodepleting chemotherapy with cyclophosphamide and fludara starting day -7. On day -2 patients will start treatment with Nivolumab every 2 weeks for a total of 4 doses to increase the activity of the infused TIL product.

Available evidence indicates that ACT is a safe and feasible treatment option in an increasing number of solid tumors, and that it should be tested in all cancer patients regardless of their cancer diagnosis.

ELIGIBILITY:
Only patients within the Danish Healthcare system are eligible for enrollment.

Inclusion Criteria:

* Histologically verified metastatic or locally advanced cancer diagnosis
* At least one lesion (>1 cm3) available for surgical resection
* Not candidate for standard treatment options
* Age of 18-70 years
* Performance status of 1 or 0.
* Life expectancy > 6 months
* One or more measurable parameter according to RECIST 1.1.
* No significant toxicity from previous cancer treatments (CTC≤1). Except alopecia (CTC≤2) or neuropathy (CTC≤2)
* Sufficient organ function, including:
* Absolute neutrophil count (ANC) ≥ 1.500 /µl
* Leucocyte count ≥ normal limit
* Platelets ≥ 100.000 /µl and <700.000 /µl
* Hemoglobin ≥ 6,0 mmol/l (regardless of prior transfusion)
* S-creatinine < 140
* S-bilirubin ≤ 1,5 times upper normal limit
* ASAT/ALAT ≤ 2,5 times upper normal limit
* Alkaline phosphatase ≤ 5 times upper normal limit
* Lactate dehydrogenase (LDH) ≤ 5 times upper normal limit
* Sufficient coagulation: PP-time>40 and INR<1,5
* Women in the fertile age must use effective contraception. This applies from inclusion and until 6 months after treatment. Birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch are all considered safe contraceptives.
* Signed statement of consent after receiving oral and written study information
* Willingness to participate in the planned treatment and follow-up and capable of handling toxicities.

Exclusion Criteria:

* A history of prior malignancies. Patients treated for another malignancy can only participate if they are without signs of disease for a minimum of 3 years after last treatment.
* Primary brain tumor or verified brain metastases
* Known hypersensitivity to one of the active drugs or excipients.
* Significant medical conditions, including but not limited to severe asthma/COLD, significant cardiac disease, poorly regulated insulin dependent diabetes mellitus.
* Creatinine clearance below 70 ml/min .
* Acute or chronic infections with HIV, hepatitis, syphilis etc.
* Severe allergies or previous anaphylactic reactions.
* Active autoimmune disease, such as autoimmune neutropenia/thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, Sjögren's syndrome, sclerodermia, myasthenia gravis, goodpastures disease, addison's disease, hashimoto's thyroiditis, graves' disease etc.
* Pregnant women and women who are breastfeeding.
* Simultaneous treatment with systemic immunosuppressive drugs (including prednisolone methotrexate etc.)
* Simultaneous treatment with other experimental drugs.
* Simultaneous treatment with other systemic anti-cancer treatments.
* Patients with active or uncontrollable hypercalcemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders H Kverneland, MD, Principal Investigator — Center for Cancer Immune Therapy, Herlev Hospital; Inge Marie Svane, MD, Prof., Study Director — Center for Cancer Immune Therapy, Herlev Hospital
Locations (1):
- Center for Cancer immune Therapy (CCIT), Dept. of Hematology and dept. of Oncology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kverneland AH, Chamberlain CA, Borch TH, Nielsen M, Mork SK, Kjeldsen JW, Lorentzen CL, Jorgensen LP, Riis LB, Yde CW, Met O, Donia M, Svane IM. Adoptive cell therapy with tumor-infiltrating lymphocytes supported by checkpoint inhibition across multiple solid cancer types. J Immunother Cancer. 2021 Oct;9(10):e003499. doi: 10.1136/jitc-2021-003499. PMID 34607899

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Autologous tumor-infiltrating lymphocytes: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion.
  Ipilimumab: One treatment with ipilimumab (3 mg/kg) prior to tumor resection.
  Nivolumab: 4 doses of nivolumab. Starting 2 days prior to TIL infusion and every 2 weeks hereafter.
  proleukin: 2 MIE s.c. injection, after TIL infusion and continuing for 2 weeks
  Cyclophosphamide: 2 doses (60 mg/kg) prior to TIL infusion
  Fludara: 5 doses (25 mg/m2) prior to TIL infusion
Period: Overall Study
Arm/Group | All Participants
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who received TIL therapy
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants and Type of Reported Adverse Events
Description: Determine the safety of the administration of TIL therapy including checkpoint inhibitors, lymphodepleting chemotherapy and Interleukin-2 for patients with cancer by reporting grade >2 adverse events according to CTCAE v. 4.0
Time Frame: Up to 2,5 years from begin of study
Population: Patients who received TIL therapy
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 25
Participants
  Neutropenia | 25
  Trombocytopenia | 22
  Anemia | 22
  Infection | 6
  Hyponatremia | 2
  Hemorrhagic cystitis | 1
  Fatique | 6
  Vertigo | 1
  Performance status drop | 4
  Thrombosis | 1
  Fever | 16
  Dyspnea | 6
  Hepatitis | 2
  Colitis | 2
  Transaminase elevation | 2
  Vomiting | 2
  Hallucination | 1
  Elevated creatinine | 1

2. Secondary Outcome: Time to Disease Progression
Description: Days of follow-up from TIL infusion until progressive cancer disease, end of follow-up or death.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Until study completion
Measure: Median (Full Range); unit: Days
Groups:
- Treated Participants: Autologous tumor-infiltrating lymphocytes: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion.
  Ipilimumab: One treatment with ipilimumab (3 mg/kg) prior to tumor resection.
  Nivolumab: 4 doses of nivolumab. Starting 2 days prior to TIL infusion and every 2 weeks hereafter.
  proleukin: 2 MIE s.c. injection, after TIL infusion and continuing for 2 weeks
  Cyclophosphamide: 2 doses (60 mg/kg) prior to TIL infusion
  Fludara: 5 doses (25 mg/m2) prior to TIL infusion
Arm/Group | Treated Participants
Number analyzed (Participants) | 25
Days | 89 [12 to 211]

3. Secondary Outcome: Overall Survival
Description: Duration of survival measured in days after adoptive cell therapy until death or end of follow-up/censoring.
Time Frame: Until study completion
Measure: Median (Full Range); unit: Days
Arm/Group | Treated Participants
Number analyzed (Participants) | 25
Days | 227 [50 to 870]

4. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CAT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: The patients were evaluated every 6-12 weeks (median 90 days) and after therapy and until study completion (max 220 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Participants
Number analyzed (Participants) | 25
Participants | 2

ADVERSE EVENTS:
Time Frame: The data was collected throughout the duration of the clinical trial. From October 2017 and until study Completion in july, 2020. For the individual patient, the reporting started at the study enrolment and ended with study exclusion but with a minimum of 6 months follow-up after the adoptive cell therapy or until study completion. Information on adverse events were collected every 6 weeks for the first 3 months and every 3 months hereafter.
Description: Patients were routinely screening for anticipated adverse events. The screening was performed every 6 weeks until the first 3 months and hereafter every 3 months for up to 2.5 years.
Arm/Group | Treated Participants
All-Cause Mortality (participants affected / at risk) | 23/25
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Participants (N=25)
Elevated bilirubin (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Refractory trombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Chylos (Skin and subcutaneous tissue disorders) | 1 (1) — After removal from lymph node
Neutropenic fever (Infections and infestations) | 1 (2)
Thrombosis in central katheter (Blood and lymphatic system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3) — Mediated by checkpoint inhibitors
Addisions crisis (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection unknown focus (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Participants (N=25)
Neutropenia (Blood and lymphatic system disorders) | 25 (28)
Trombocytopenia (Blood and lymphatic system disorders) | 23
Anemia (Blood and lymphatic system disorders) | 22 (28)
Fatigue (General disorders) | 20 (20)
Nausea (General disorders) | 24 (24)
Vomiting (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 10
Obstipation (Gastrointestinal disorders) | 6
Oral mucositis (Infections and infestations) | 14 (23)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 8 (10)
Febrile neutropenia (General disorders) | 23 (25)
Edema (Skin and subcutaneous tissue disorders) | 3 (3)
Elevated liver enzymes (Hepatobiliary disorders) | 4 (4)
Infections (Infections and infestations) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (8)
Granuloma (Skin and subcutaneous tissue disorders) | 5 (5)
Muscle/joint pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Hallucinations (Psychiatric disorders) | 4 (4)
Vertigo (Nervous system disorders) | 2 (2)
Hyponatremia (Renal and urinary disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Autoimmune reactions (Immune system disorders) | 6 (8)
Fever (General disorders) | 18 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03296137/Prot_SAP_000.pdf